CLINICAL TRIAL: NCT07325149
Title: Exoskeletal-assisted Walking Combined With Transcutaneous Spinal Cord Stimulation: Effect on Imaging and Serum Biomarkers of Skeletal Muscle Mass and Bone Strength.
Brief Title: The Effect of Exoskeletal-assisted Walking Combined With Transcutaneous Spinal Cord Stimulation on Bone Strength.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bronx VA Medical Center (U.S. Federal Agency)
Collaborators: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Christopher M. Cirnigliaro, Investigator, Research Health Science Specialist, Bronx VA Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1914010-2; IK2 RD000484-01A1 (Other Grant/Funding Number: Department of Veterans Affairs Rehabilitation Research, and Development Translation)
Record Dates: First submitted 2025-12-18; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Secondary Osteoporosis; Sarcopenia
Keywords: Spinal Cord Injury; Transcutaneous Spinal Cord Stimulation; Bone Mineral Density; Exoskeleton-Assisted Walking; Muscle Cross Sectional Area
MeSH Terms: conditions — Sarcopenia; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Exoskeleton-Assisted Walking (EAW) + active Transcutaneous Spinal Cord Stimulation (tSCS) (Experimental): The EAW + active tSCS group will receive simultaneous lumbosacral tSCS while simultaneously performing EAW.
  Interventions: Device: Exoskeleton-Assisted Walking (EAW) + active Transcutaneous Spinal Cord Stimulation (tSCS)
- Exoskeleton-assisted walking (EAW) + sham Transcutaneous Spinal Cord Stimulation (tSCS) (Sham Comparator): The EAW + sham tSCS group will receive simultaneous lumbosacral sham tSCS while simultaneously performing EAW. Participants in both groups will receive 60 minutes of EAW + sham tSCS overground training per session for a total of 108 sessions (3 X week for 36 weeks).
  Interventions: Device: Exoskeleton-assisted walking (EAW) + sham Transcutaneous Spinal Cord Stimulation (tSCS)

INTERVENTIONS:
Device: Exoskeleton-Assisted Walking (EAW) + active Transcutaneous Spinal Cord Stimulation (tSCS) — The full electrical signal is delivered during lumbosacaral tSCS treatment while simultaneously performing EAW. Participants in both groups will receive 60 minutes of EAW + active tSCS overground training per session for a total of 108 sessions (3 X week for 36 weeks).
  Arms: Exoskeleton-Assisted Walking (EAW) + active Transcutaneous Spinal Cord Stimulation (tSCS)
Device: Exoskeleton-assisted walking (EAW) + sham Transcutaneous Spinal Cord Stimulation (tSCS) — The lumbosacral tSCS electrical signal is set too low to have any biological effect while simultaneously performing EAW.
  Arms: Exoskeleton-assisted walking (EAW) + sham Transcutaneous Spinal Cord Stimulation (tSCS)

SUMMARY:
Immobilization following spinal cord injury (SCI) results in muscle and bone loss below the level of injury, which ultimately predisposes to fracture at several sites throughout the legs and can lead to several medical complications that can devastate quality of life. There is a scarcity of research that has successfully implemented rehabilitation and/or exercise training interventions to preserve the musculoskeletal system during the acute phase SCI, or possibly reverse the muscle and bone loss that has already occurred in chronic SCI. This study will compare the effect of exoskeleton-assisted walking (EAW) training combined with transcutaneous spinal cord stimulation (tSCS) (EAW + active tSCS), to that of EAW + sham tSCS, on measures of muscle and bone health in a cohort of chronically injured motor incomplete SCI. A successful outcome would expand treatment options to improve musculoskeletal health over the lifetime.

DETAILED DESCRIPTION:
Background: Immobilization results in bone loss that predisposes to osteoporosis and fracture, which may be complicated by non-union, infection, and deep venous thrombosis. Reduced muscular contraction after SCI and the elevated release of cortisol contribute to a catabolic state, resulting in a loss of lean tissue mass (LTM) below the level of lesion. Six months after motor-complete SCI, the average muscle cross-sectional area (CSA) significantly decreases at the quadriceps, hamstrings, and hip adductors (14-16%), and 12% and 24% at the soleus and gastrocnemius, respectively. Following SCI, the quadricep muscles generate less total force and force per unit area when evoked by surface electrode electrical stimulation. This loss of muscle CSA and strength in the lower extremities limits the ability to stand, ambulate, and preserve bone - even if neural regenerative strategies could be implemented in the future. In addition to the marked skeletal muscle atrophy, persons with non-ambulatory motor-complete SCI also experience a precipitous loss of bone mineral content (BMC) and bone mineral density (BMD) by as much as 1% per week below the level of lesion. In individuals with motor-incomplete lesions who have not reached their ambulatory potential, there is still considerable bone loss due to immobilization that can reach the fracture threshold years after injury. This rapid bone loss during the first two years after SCI results in volumetric BMD (vBMD) at the DF and PT decreasing by ~ 50% and 26% at the trabecular and cortical compartments, respectively. During the chronic phase of SCI bone loss continues more slowly throughout the individuals lifetime. This loss in muscle and bone places individuals with SCI at high risk for fragility fracture. More than 50% of individuals with SCI experience a fragility fracture over the course of their lifetimes.

Objectives: Aim 1: To compare the effects of 108 sessions of EAW + sham tSCS versus EAW + active tSCS on the muscle-bone unit in wheelchair-dependent chronic SCI participants.

Aim 2 (exploratory): To determine the acute time-course responses for serum/plasma biomarkers of bone resorption and formation, muscle contractile activity, and the mRNA profiles of circulating exosomes collected prior to (time 0), and again 30, 60, 120, 180, minutes and 24, and 48 hours following an acute session of both the EAW + active tSCS and EAW + sham tSCS training interventions.

Setting: Participant enrollment, the clinical trial intervention (EAW + sham tSCS versus EAW + active tSCS), EMG data collection, dual energy X-ray absorptiometry (DXA), peripheral quantitative computed tomography (pQCT), magnetic resonance imaging (MRI) to measure the cross-sectional area of the mid-thigh, and the time-course responses for serum/plasma biomarkers of bone resorption and formation and muscle contractile activity will be performed at the Kessler Foundation and the James J. Peters VA Medical Center.

Design: After meeting eligibility criteria, wheelchair users with chronic SCI will be block randomized into the EAW + active tSCS group or the EAW + sham tSCS group (n=12 in each group). Both groups will receive 60 minutes of EAW overground training per session for a total of 108 sessions (3 X week for 36 weeks). In addition to the EAW training, the EAW + active tSCS group will receive simultaneous lumbosacral tSCS targeted to activate the locomotor central pattern generator.

Participants: Twenty-four participants (12 participants/group) with SCI will be recruited over a 4-year period and randomly assigned to an EAW + sham tSCS or EAW + active tSCS group. At the end of the first year, approximately 3 participants will have completed the protocol.

Outcome measures: At baseline, the investigators will perform imaging to measure bone density and strength, surface EMG to assess muscle contractility, and a time-course response for serum muscle and bone biomarkers following an acute bout of EAW. The investigators will capture these same data again after ~54 training sessions (mid-point), and after 108 training sessions (month 9 timepoint). In addition, MRI of both legs for muscle CSA will be performed at the baseline and month 9 time point.

ELIGIBILITY:
* Participant Screening:

  1. International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) neurological assessment examination to determine the level and completeness of SCI when participants screen for entry into the study. The ISNCSCI exam will be performed by the study physician using a tool that assesses sensory function (light touch and pinprick) in each dermatome (A dermatome is an area of skin that sends touch, pain, temperature, and other sensory signals back to the brain) and motor function (motor function is a general term to describe the way muscles create movement) in ten key muscles. This test will determine the level of SCI, defined as the lowest spinal level with normal function, and assigns a classification of severity according to the ISNCSCI scale. In this study, both ISNCSCI grade C and grade D would make a participant eligible for this study.
  2. DXA study to assess bone mineral density (BMD) at the total hip (TH), distal femur (DF), and proximal tibia (PT) that will be compared to the cutoff values described in the exclusion criteria section.
  3. Medical history and exam to ensure medical health, anthropometric compatibility for EAW, and to identify fragility or traumatic fractures, unhealed fractures, and signs of swelling, bruising, and discoloration of the legs.
* Inclusion Criteria:

  1. Between the ages of 21-60 years old
  2. Non-walkers with an SCI greater than 3 years post injury.
  3. As measured by a member of the study staff, participants who have a lower extremity motor score greater or equal to 16 on the INSCSCI exam with an impairment grade of C or D.
  4. Neurologic level of injury as determined by study staff between C5-T10 (completed at participant's screening).
  5. Capable of gripping Lofstrand crutches and/or a walker without assistance.
  6. Wheelchair reliant 100% of the time.
  7. Height is between 62 inches and 74 inches.
  8. Weight less than 220lbs.
  9. Anthropometric compatibility with the EAW device:

     * Thigh length between 14 and 19 in (36 and 48 cm).
     * Shank length between 17 and 22 in (43 and 55 cm).
* Exclusion Criteria:

  1. As determined by the study physician from the screening health exam, a history of fragility or traumatic fractures, unhealed fractures, and signs of swelling, bruising, and discoloration of the legs.
  2. Current bone disease diagnosis (e.g., osteomyelitis, hyperparathyroidism)
  3. As determined by the study physician from the screening DXA study, a T-score at the total hip < -3.5 or aBMD of the knee (proximal tibia and/or distal femur) < 0.60 g/cm2 from the DXA screen
  4. Positive pregnancy test at any of the study intervention or assessment visits, or if female participants plan to become pregnant over the course of the study, they will be excluded or withdrawn (if already enrolled) from participation.
  5. Currently in a gym/rehabilitation program performing ambulatory interventions such as EAW, as determined by the study staff.
  6. Currently prescribed any medications that can affect muscle and/or bone metabolism, as determined by the study staff.

Exclusion Criteria from MRI Safety Screening:

1. Medically unsafe to receive an MRI scan.
2. Claustrophobia
3. Baclofen pump
4. Body metal, including any of the following:

   * metal fragments or pieces in eyes or any other part of body
   * pacemakers or other implanted electrical devices
   * aneurysm clips (metal clips on wall of a large artery)
   * metallic prostheses (metal pins and heart valves)
   * internal hearing aids (cochlear implants)
   * permanent eyeliner
   * shrapnel fragments
   * piercing that cannot be removed

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-07-01 (Estimated); Primary Completion 2031-06-30 (Estimated); Study Completion 2033-06-01 (Estimated)

PRIMARY OUTCOMES:
Muscle cross sectional area of the mid-thigh | Obtained prior to starting the study at enrollment (baseline) and again after 9 months of participating in the study interventions.
  EAW + active tSCS will increase muscle cross sectional area of the mid-thigh more than EAW + sham tSCS.

OTHER OUTCOMES:
Bone Strength at the Distal Femur and Proximal Tibia | Obtained prior to starting the study at enrollment (baseline), after ~54 training sessions (4.5 months), with a final measurement completed after 9 months of the training interventions.
  EAW + active tSCS will increase bone strength at the distal femur and proximal tibia more than EAW + sham tSCS.
Muscle and Bone Serum and Plasma Biomarker Time-Course Response | Obtained prior to starting the study at enrollment (baseline), after ~54 training sessions (4.5 months), with a final measurement completed after 9 months of the training interventions.
  An intravenous line will be placed to draw serial serum and plasma samples prior to (time 0), and again 30, 60, 120, 180, minutes and 24, and 48 hours following an acute session of either an EAW + sham tSCS or an EAW + active tSCS training intervention depending on that participant's group assignment.
Seated and Supine Electromyography (EMG) assessments of Muscle Activation | Obtained prior to starting the study at enrollment (baseline), after ~54 training sessions (4.5 months), with a final measurement completed after 9 months of the training interventions.
  Surface EMG data will be collected from muscles in each leg to assess surface EMG amplitudes of these muscles during attempts at volitional knee extension and flexion and ankle plantar- and dorsi-flexion using surface sensors. Furthermore, the resting EMG protocol will be performed to determine the individualized mapping to determine the minimum tSCS intensity required to evoke a motor evoked potential (MEP).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher P Cardozo, M.D., Study Director — James J. Peters VA Medical Center
Locations (1):
- Kessler Foundation, West Orange, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
At this time, the investigators must declare that IPD will not be shared with other investigators, as the VA has not approved a plan and is currently not in place at our VA research laboratory. The investigators anticipate a policy will be approved over the next 24 months to share IPD with other investigators. Once an approved plan is in place, it will be added to the study protocol and the PRS site for this trial.

REFERENCES:
- [Result] Totosy de Zepetnek JO, Craven BC, Giangregorio LM. An evaluation of the muscle-bone unit theory among individuals with chronic spinal cord injury. Spinal Cord. 2012 Feb;50(2):147-52. doi: 10.1038/sc.2011.99. Epub 2011 Sep 6. PMID 21894164
- [Result] Samejima S, Caskey CD, Inanici F, Shrivastav SR, Brighton LN, Pradarelli J, Martinez V, Steele KM, Saigal R, Moritz CT. Multisite Transcutaneous Spinal Stimulation for Walking and Autonomic Recovery in Motor-Incomplete Tetraplegia: A Single-Subject Design. Phys Ther. 2022 Jan 1;102(1):pzab228. doi: 10.1093/ptj/pzab228. PMID 35076067
- [Result] Gerasimenko Y, Gorodnichev R, Moshonkina T, Sayenko D, Gad P, Reggie Edgerton V. Transcutaneous electrical spinal-cord stimulation in humans. Ann Phys Rehabil Med. 2015 Sep;58(4):225-231. doi: 10.1016/j.rehab.2015.05.003. Epub 2015 Jul 20. PMID 26205686
- [Result] Gerasimenko YP, Lu DC, Modaber M, Zdunowski S, Gad P, Sayenko DG, Morikawa E, Haakana P, Ferguson AR, Roy RR, Edgerton VR. Noninvasive Reactivation of Motor Descending Control after Paralysis. J Neurotrauma. 2015 Dec 15;32(24):1968-80. doi: 10.1089/neu.2015.4008. Epub 2015 Aug 20. PMID 26077679
- [Result] Karelis AD, Carvalho LP, Castillo MJ, Gagnon DH, Aubertin-Leheudre M. Effect on body composition and bone mineral density of walking with a robotic exoskeleton in adults with chronic spinal cord injury. J Rehabil Med. 2017 Jan 19;49(1):84-87. doi: 10.2340/16501977-2173. PMID 27973679
- [Result] Shackleton C, Evans R, West S, Derman W, Albertus Y. Robotic Walking to Mitigate Bone Mineral Density Decline and Adverse Body Composition in Individuals With Incomplete Spinal Cord Injury: A Pilot Randomized Clinical Trial. Am J Phys Med Rehabil. 2022 Oct 1;101(10):931-936. doi: 10.1097/PHM.0000000000001937. Epub 2021 Dec 6. PMID 34864766